CLINICAL TRIAL: NCT03052985
Title: Observatory of Materiovigilance After Surgery of Urinary Incontinence or Prolapse in Women.
Brief Title: Materiovigilance After Urinary Incontinence or Prolapse Surgery
Acronym: VIGI-MESH
Status: Active, not recruiting | Type: Observational
Sponsor: Poitiers University Hospital (Other)
Collaborators: Agence Nationale de sécurité du Médicament (Other)
Responsible Party: Sponsor
Other Study IDs: 2016-A01868-43
Record Dates: First submitted 2017-02-10; First posted 2017-02-14 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Pelvic Organ Prolapse; Rectal Prolapse; Urinary Stress Incontinence
Keywords: medical devices (meshes); surgery
MeSH Terms: conditions — Pelvic Organ Prolapse; Rectal Prolapse; Urinary Incontinence, Stress

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: urinary incontinence, pelvic organ or rectal prolapse surgery — The observatory is planned for following women after surgery for urinary incontinence, pelvic organ prolapse, or rectal prolapse whatever the type of surgery (by laparoscopy, laparotomy or vginal route) or the use of a mesh

SUMMARY:
Observatory of Materiovigilance After Surgery of Urinary Incontinence or Prolapse in Women Implantable medical devices (meshes) used in pelvic organ prolapse surgery (genital prolapse, rectal prolapse), or incontinence surgery may be source of severe complications.

DETAILED DESCRIPTION:
RATIONAL Implantable medical devices (meshes) used in pelvic organ prolapse surgery (genital prolapse, rectal prolapse), or incontinence surgery may be source of severe complications.

MAIN OBJECTIVE Estimate the incidence of severe complications during or after surgery of urinary incontinence or pelvic organ prolapse in adult women depending on the type of surgery performed.

SECONDARY OBJECTIVES Estimate the incidence of severe complications after urinary incontinence or prolapse surgery as a function of time since surgery.

Compare the incidence rates of severe complications considering the type of procedure (with or without mesh, vaginal or laparoscopic, etc.), comorbidities, mesh type, surgeon experience, and surgical volume centre.

Report the health and satisfaction of operated women. Estimate the risk of revision surgery for failure or recurrence.

MAIN OUTCOME Per- and post-operative complications (less than 12 months after surgery), or late (after 12 months) severe (grade III or higher according to the Clavien-Dindo classification)

OTHER OUTCOMES Time lapse of occurrence of severe complications Surgical recovery for failure or recurrence Health and perceived improvement (OMS, EQ5D, an PGI-I questionnaires)

DESIGN Prospective multicentre cohort allowing the constitution and analysis of an observatory off surgery for genital prolapse, rectal prolapse and urinary stress incontinence in women.

INCLUSION CRITERIA

* Operated for urinary incontinence, genital prolapse, or rectal prolapse in one of the centres participating in the observatory
* 18 years old or more.

SUBJECTS NUMBER Estimated at 3000 per year during 5 years in 18 participating centres

STUDY LENGTH Duration of the inclusion period: 2 years with the initial grant from ANSM (Agence Nationale de Sécurité du Médicament et des produits de santé, French Medicines and Healthcare Products Regulatory Agency), after new funding by ANSM 5 years of inclusion in total.

Duration of participation of subjects: 2 years with grant from ANSM, after the new funding by ANSM 10 years.

Total duration of the study: 3 years with the grant from ANSM, 15 years with the new funding.

ANALYSIS PLANNED The one-year analysis will be based on multivariate logistic regression analysis (considering confounding factors). The 10-year (or intermediate-term) analysis will use survival analysis methods to account for delays in complications: Kaplan-Meier curves; Model of Cox proportional hazards.

PERSPECTIVES The observatory should make it possible to precise the tolerance and the short- and long-term consequences of the use of these implantable devices (meshes) in pelvic organ prolapse or incontinence surgery in women and to specify the risk factors for severe complications.

The observatory will enable to make comparisons between the different types of meshes and different surgical procedures, and to identify those that may present problems.

Clinical practice recommendations may be issued as well as standards for marketing.

ELIGIBILITY:
Inclusion Criteria:

* Operated for urinary incontinence, pelvic organ prolapse, or rectal prolapse in one of the centres participating in the observatory
* 18 years old or more.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women operated for urinary incontinence, pelvic organ prolapse, or rectal prolapse in one of the centres participating in the observatory, aged 18 years old or more.
Sampling Method: Non-Probability Sample
Enrollment: 19000 (Actual)
Dates: Start 2017-02-14 (Actual); Primary Completion 2033-05-01 (Estimated); Study Completion 2033-05-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of severe complications | 10 years
  Grade III or more according to Clavien-Dindo classification

SECONDARY OUTCOMES:
Time lapse of occurrence of severe complications | 10 years
Surgical recovery for failure or recurrence | 10 years
  Number participent with new revision surgery for failure Number participent with new revision surgery for recurrence
Health and perceived improvement | 10 years
  Scale OMS/ ECOG Eastern Cooperative Oncology Groupone covers six values, from 0 to 5, where 0 represents a good state of health and 5 the death.
Health and perceived improvement | 10 years
  EQ5D is a standardised measure of health status developed
  Each of the 5 dimensions comprising the EQ-5D descriptive system is divided into 5 levels of perceived problems :
  * Level 1 : indicating no problem
  * Level 2 : indicating slight problems
  * Level 3 : indicating moderate problems
  * Level 4 : indicating severe problems
  * Level 5 : indicating extreme problems
Health and perceived improvement | 10 years
  PGI-I, Patient Global Impression of Improvement, is a transition scale that is a single question asking the patient to rate their urinary tract condition now, as compared with how it was prior to before beginning treatment on a scale from 1. Very much better to 7. Very much worse.

CONTACTS AND LOCATIONS:
Overall Officials: Xavier FRITEL, PhD, MD, Principal Investigator — Poitiers University Hospital
Locations (31):
- France (31):
  - Centre l'Avancée - Clinique Axium, Aix-en-Provence
  - C.H.U. d'Angers, Angers
  - CHRU de Besançon, Besançon
  - Centre Hospitalier de Béthune, Béthune
  - CHU de Bordeaux, Bordeaux
  - CHU Caen, Caen
  - Centre Hospitalier Camille Guérin, Châtellerault
  - Hôpital Antoine-Béclère, Clamart
  - Chu Estaing, Clermont-Ferrand
  - Centre Hospitalier de Dunkerque, Dunkirk
  - Polyclinique d'Hénin-Beaumont, Hénin-Beaumont
  - Hopital La Rochelle- Ré- Aunis, La Rochelle
  - CHU Lille, Lille
  - Hôpital St Vincent De Paul, Lille
  - CHU de Limoges, Limoges
  - Hospices Civils de Lyon, Lyon
  - Clinique BEAUSOLEIL, Montpellier
  - CHRU de NANCY, Nancy
  - CHU Nantes, Nantes
  - CHRU Carémeau, Nîmes
  - La Pitié-Salpêtrière, Paris
  - Hôpital Bichat, Paris
  - Groupe Hospitalier Diaconesses Croix Saint-Simon, Paris
  - Centre briochin d'Urologie, Plérin
  - CHI Poissy-St-Germain, Poissy
  - CHU de Poitiers, Poitiers
  - CHU de Reims, Reims
  - CHU Strasbourg, Strasbourg
  - Hopital Foch, Suresnes
  - Clinique UROVAR, Toulon
  - CHU de Toulouse, Toulouse

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Carter E, Johnson EE, Still M, Al-Assaf AS, Bryant A, Aluko P, Jeffery ST, Nambiar A. Single-incision sling operations for urinary incontinence in women. Cochrane Database Syst Rev. 2023 Oct 27;10(10):CD008709. doi: 10.1002/14651858.CD008709.pub4. PMID 37888839